CLINICAL TRIAL: NCT06380452
Title: Phase III Multicenter, Prospective, Randomized, Double-blind Study Comparing the Efficacy and Safety of Therapy for Scabies With Two Differently Concentrated Permethrin Creams.
Brief Title: Therapy for Scabies With Two Differently Concentrated Permethrin Creams
Acronym: SKABUP
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Infectopharm Arzneimittel GmbH (Industry)
Collaborators: Winicker Norimed GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SKABUP; 2023-507925-41-00 (Other: EU-Trial-Nr. (EMA))
Record Dates: First submitted 2024-04-16; First posted 2024-04-23 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Scabies
MeSH Terms: conditions — Scabies

STUDY DESIGN:
Intervention Model Description: The SKABUP study is a prospective, randomized, double-blind, 2-arm superiority study in a group sequential design with recruitment stop and interim analysis after 172 patients. If there is no evidence of superiority in the interim analysis, the study will be continued unchanged up to the planned number of 220 patients and will be terminated and analyzed regularly.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 5% Permethrin Creme (Active Comparator): Permethrin Cream 5 % is the already approved standard therapeutic agent InfectoScab 5 % Cream, contains the active ingredient permethrin in a 5 % concentration and is used for the topical treatment of scabies. The cream is also used as a topical cream, e.g. after washing hands.
  Interventions: Drug: 5% Permethrin Creme
- 10% Permethrin Creme (Experimental): Permethrin Cream 10 % also contains the active ingredient permethrin, but in double the concentration, and otherwise corresponds to the approved standard therapeutic agent InfectoScab 5 % Cream in terms of the main other ingredients. This is also used for the topical treatment of scabies, as well as for re-creaming, e.g. after washing hands.
  Interventions: Drug: 10% Permethrin Creme

INTERVENTIONS:
Drug: 5% Permethrin Creme — At visit V0, the investigational cream is applied once topically to the whole body. For patients who are not cured at visit V1, i.e. 14 days later, the application is repeated analogously once at this time.
  Arms: 5% Permethrin Creme
Drug: 10% Permethrin Creme — At visit V0, the investigational cream is applied once topically to the whole body. For patients who are not cured at visit V1, i.e. 14 days later, the application is repeated analogously once at this time.
  Arms: 10% Permethrin Creme

SUMMARY:
The multi-center, prospective, randomized, double-blind phase III clinical trial will primarily investigate the efficacy and safety of treatment of scabies with Permethrin Cream 5% (approved drug InfectoScab 5% Cream) in direct comparison with Permethrin Cream 10%.

The trial participants will be randomly assigned and blinded to either Permethrin Cream 5% or Permethrin Cream 10%.

DETAILED DESCRIPTION:
The SKABUP study is a multi-center, prospective, randomized, double-blind phase III clinical trial. The aim of this SKABUP study is to compare the efficacy and safety of topical therapy with permethrin 5% and permethrin 10% in a multicenter randomized double-blind setting in order to demonstrate the possible superiority of the 10% permethrin cream over the current standard therapy with permethrin 5% cream. In order to demonstrate a possible difference in efficacy as clearly as possible, the study will be conducted in dermatology clinics and without extensive exclusion of previous therapies in the patient's medical history.

The primary objective of the SKABUP study is the clincal efficacy (therapeutic success yes/no) after completion of treatment (one or - if necessary - two applications), i.e. treatment success on day 14 (for study participants with only one application of investigational product) or on day 28 (for study participants with repeated application of investigational product).

A total of 220 scabies patients aged between 2 and 85 years are to be included in the study (clinical trial). After 172 patients, however, recruitment will be stopped and an interim evaluation carried out. If there is proof of superiority, the study will be terminated; if there is no proof of superiority, it will be continued unchanged. Study drop-outs, i.e. patients included in the study with at least one application of an investigational product whose participation in the study ends prematurely, will not be replaced.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed acute scabies disease: Detection of mites and/or mite nymphs and/or mite larvae, by reflected light microscopy or light microscopy of skin samples, at scabies-typical predilection sites
* Age between 2 years and 85 years
* Written informed consent of the study participant (if of legal age) or all legal guardians (for underage study participants < 12 years) or all legal guardians and the study participant (for underage study participants ≥ 12 years)
* Practicable application of the trial medication by trained specialist staff at the trial site

Exclusion Criteria:

* Pre-treatment with antiscabiosa in the last 14 days
* Combined antiscabial treatment (i.e. simultaneous/simultaneous topical and systemic scabies treatment with medication) in the last 3 months
* Known intolerance to permethrin, other pyrethroids, chrysanthemums or any of the other ingredients of the study medication
* Scabies crustosa
* Impetiginization/eczematization requiring inpatient treatment
* Body weight > 120 kg
* Pregnancy, breastfeeding
* Clinically relevant immunodeficiency (of any kind, including extensive local therapy (>20% body surface) with corticosteroids > 2 weeks in the last 4 weeks or ≥ 10 mg prednisolone equivalent >7 days in the last 4 weeks - even without signs of scabies crustosa)
* Other serious illnesses which, in the opinion of the investigator, prevent the patient from participating in the study
* Planned systemic use of corticosteroids
* Planned or previous (last 4 weeks) use of systemic or cutaneous non-steroidal immunosuppressants
* Apparent unreliability or unwillingness to cooperate
* Inability to understand and comply with study instructions
* Known alcohol, medication or drug dependence
* Placement in a facility where people live together for long periods of time, are cared for or receive medical care, and where close skin-to-skin contact is common, or placement in an institution ordered by a court/authority
* 5 or more close contacts (persons with close, extensive skin-to-skin contact with the scabies patient for more than 5-10 minutes)
* Close contact person who refuses scabies treatment or for whom treatment is not possible
* Dependence on sponsor or investigator
* Previous participation in a clinical trial in the last 30 days or in the same clinical trial

Ages: 2 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
clinical efficacy (yes/no) | day 14 - day 28
  The primary outcome criterion is defined as clinical efficacy (therapeutic success yes/no) after completion of treatment (one or - if necessary - two applications) i.e. treatment success on day 14 (for study participants with only one investigational product application) or on day 28 (for study participants with repeated investigational product application).

SECONDARY OUTCOMES:
effectiveness at Visit 1 | day 14
  therapy success at Visit 1
frequency of therapy success | day 0 - day 28
  frequency of therapy success after only one application in relation to the overall frequency of therapy success (after completion of treatment)
itching | day 0 - day 28
  itching (Numerical Rating Scale (NRS) from 0-10) and change in itching vs. baseline (scale differences) for all visits
patients with evidence of mites | day 0 - day 28
  proportion of patients (in %) with evidence of mites (incl. nymphs and larvae, reflected light microscopy or light microscopy of skin samples) for all visits
patients with use of antiscabiosa not compliant with the protocol | day 0 - day 28
  proportion of patients with use of antiscabiosa not compliant with the study protocol for all visits
patients with new scabies efflorescences | day 0 - day 28
  Proportion of patients with new scabies efflorescences for all visits
patients with "additional confirmed" treatment failure | day 0 - day 28
  patients with "additional confirmed" treatment failure (in %): Proportion of patients with new scabies efflorescences at the end of treatment OR with mite detection by microscopic examination of a skin sample OR use of other antiscabio-sa not conforming to the study protocol
AEs, SAEs, ADRs, SUAWs | day 0 - day 28
  AEs, SAEs, ADRs, SUAWs (total frequency, type, severity, causality, with frequencies, with separate presentation of local reactions)

CONTACTS AND LOCATIONS:
Overall Officials: Cord Sunderkötter, Prof. Dr., Study Director — Universitätsklinik und Poliklinik für Dermatologie une Venerologie, Halle (Saale)

IPD SHARING:
Plan to Share IPD: No